CLINICAL TRIAL: NCT00732160
Title: Aldosterone and Glucose Homeostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Matt Luther, Assistant Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 080248
Record Dates: First submitted 2008-08-05; First posted 2008-08-11 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose; Insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HS-V/A; LS-V/A (Experimental): High Sodium diet- Vehicle infusion then Aldosterone infusion Low Sodium diet- Vehicle infusion then Aldosterone infusion
  Interventions: Drug: Aldosterone infusion (A); Drug: Vehicle Infusion (V); Other: High Sodium Diet (HS); Other: Low Sodium Diet (LS)
- HS-A/V; LS-A/V (Experimental): High Sodium diet- Aldosterone infusion then Vehicle infusion Low Sodium diet- Aldosterone infusion then Vehicle infusion
  Interventions: Drug: Aldosterone infusion (A); Drug: Vehicle Infusion (V); Other: High Sodium Diet (HS); Other: Low Sodium Diet (LS)
- LS-V/A; HS-V/A (Experimental): Low Sodium diet- Vehicle infusion then Aldosterone infusion High Sodium diet- Vehicle infusion then Aldosterone infusion
  Interventions: Drug: Aldosterone infusion (A); Drug: Vehicle Infusion (V); Other: High Sodium Diet (HS); Other: Low Sodium Diet (LS)
- LS-A/V; HS-A/V (Experimental): Low Sodium diet- Aldosterone infusion then Vehicle infusion High Sodium diet- Aldosterone infusion then Vehicle infusion
  Interventions: Drug: Aldosterone infusion (A); Drug: Vehicle Infusion (V); Other: High Sodium Diet (HS); Other: Low Sodium Diet (LS)

INTERVENTIONS:
Drug: Aldosterone infusion (A) — Infusion of exogenous aldosterone (0.7 mcg/kg/hr for 12.5 hrs)
  Other Names: placebo
Drug: Vehicle Infusion (V) — Vehicle infusion for 12.5 hours
Other: High Sodium Diet (HS) — 160 mmol/d sodium diet for 7 days
Other: Low Sodium Diet (LS) — 20 mmol/d sodium diet for 9 days

SUMMARY:
Determine the effect of aldosterone on how the body handles glucose (sugar).

DETAILED DESCRIPTION:
Determine the effect of aldosterone on glucose metabolism in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory subjects, 18 to 70 years of age, inclusive
2. For female subjects, the following conditions must be met:

   a postmenopausal status for at least 1 year, or b status-post surgical sterilization, or c if of childbearing potential, utilization of adequate birth control and willingness to undergo urine beta-hcg testing prior to drug treatment and on every study day
3. Metabolic Syndrome as defined by the presence of > 3 of the following:

a Systolic Blood Pressure > 130 mm Hg OR Diastolic Blood Pressure > 85 mm Hg. b Glucose Intolerance (Fasting Plasma Glucose > 100 mg/dL) c Increased triglyceride level > 150mg/dL (1.7mmol/L) d Decreased levels of HDL cholesterol For males, less than 40 mg/dL For females, less than 50 mg/dL e Waist circumference For males, greater than 40 inches (102 cm) For females, greater than 35 inches (89 cm).

Exclusion Criteria:

1. Previously diagnosed Type I Diabetes , or the use of anti-diabetic medication. Subjects with type II diabetes not on medication will be allowed to participate if fasting blood glucose is <200mg/dL.
2. Prior allergies to medications used in the study protocol (e.g. L-arginine, potassium chloride).
3. Screening plasma potassium <3.5 mmol/L or use of chronic potassium supplements for the treatment of hypokalemia
4. Use of hormone replacement therapy
5. If on statin therapy for hypercholesterolemia, a change in dose within the past 6 months.
6. Breast-feeding
7. Cardiovascular disease such as prior myocardial infarction, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
8. Treatment with anticoagulants
9. History of serious neurologic disease such as cerebral hemorrhage, stroke, seizure, or transient ischemic attack
10. History or presence of immunological or hematological disorders
11. Diagnosis of asthma requiring use of inhaled beta agonist >1 time per week
12. Clinically significant gastrointestinal impairment that could interfere with drug absorption
13. Impaired hepatic function [aspartate amino transaminase (AST) and/or alanine amino transaminase (ALT) >2.0 x upper limit of normal range]
14. Impaired renal function [estimated glomerular filtration rate (eGFR) of <60ml/min] as determined by the four-variable Modification of Diet in Renal Disease (MDRD) equation, where serum creatinine (Scr) is expressed in mg/dl and age in years:
15. eGFR <60 ml/min
16. Hematocrit <35%
17. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult, such as arthritis treated with non-steroidal antiinflammatory drugs
18. Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
19. Treatment with lithium salts
20. History of alcohol or drug abuse
21. Treatment with any investigational drug in the 1 month preceding the study
22. Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
23. Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Luther, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Ramirez CE, Shuey MM, Milne GL, Gilbert K, Hui N, Yu C, Luther JM, Brown NJ. Arg287Gln variant of EPHX2 and epoxyeicosatrienoic acids are associated with insulin sensitivity in humans. Prostaglandins Other Lipid Mediat. 2014 Oct;113-115:38-44. doi: 10.1016/j.prostaglandins.2014.08.001. Epub 2014 Aug 28. PMID 25173047
- [Derived] Luther JM, Byrne LM, Yu C, Wang TJ, Brown NJ. Dietary sodium restriction decreases insulin secretion without affecting insulin sensitivity in humans. J Clin Endocrinol Metab. 2014 Oct;99(10):E1895-902. doi: 10.1210/jc.2014-2122. Epub 2014 Jul 16. PMID 25029426
- [Derived] Brown JM, Williams JS, Luther JM, Garg R, Garza AE, Pojoga LH, Ruan DT, Williams GH, Adler GK, Vaidya A. Human interventions to characterize novel relationships between the renin-angiotensin-aldosterone system and parathyroid hormone. Hypertension. 2014 Feb;63(2):273-80. doi: 10.1161/HYPERTENSIONAHA.113.01910. Epub 2013 Nov 4. PMID 24191286

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants did not start the study (5 Participants did Not Meet inclusion or exclusion criteria, 6 declined participation)
Groups:
- HS-V/A; LS-V/A: High Sodium diet- Vehicle then Aldosterone Low Sodium diet- Vehicle then Aldosterone
- HS-A/V; LS-A/V: High Sodium diet- Aldosterone then Vehicle Low Sodium diet- Aldosterone then Vehicle
- LS-V/A; HS-V/A: Low Sodium diet- Vehicle then Aldosterone High Sodium diet- Vehicle then Aldosterone
- LS-A/V; HS-A/V: Low Sodium diet- Aldosterone then Vehicle High Sodium diet- Aldosterone then Vehicle
Period: Overall Study
Arm/Group | HS-V/A; LS-V/A | HS-A/V; LS-A/V | LS-V/A; HS-V/A | LS-A/V; HS-A/V
Started | 7 | 5 | 6 | 5
HS Vehicle | 7 | 5 | 3 | 3
HS Aldosterone | 7 | 5 | 3 | 3
LS Vehicle | 2 | 1 | 6 | 5
LS Aldosterone | 2 | 1 | 6 | 5
Completed | 2 | 1 | 3 | 3
Not Completed | 5 | 4 | 3 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — scheduling | 4 | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Healthy volunteers
Groups:
- Total: Total of all reporting groups
Arm/Group | HS-V/A; LS-V/A | HS-A/V; LS-A/V | LS-V/A; HS-V/A | LS-A/V; HS-A/V | Total
Number analyzed (Participants) | 7 | 5 | 6 | 5 | 23
Age, Continuous [Mean (Full Range); unit: years] | 25.1 [21.7 to 30.1] | 29.2 [24.5 to 36.5] | 32.5 [20.9 to 47.5] | 27.2 [20.8 to 30.8] | 28.4 [20.8 to 47.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 2 | 11
  Male | 4 | 2 | 3 | 3 | 12
Glucose (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 85.3 (7.6) | 85.4 (7.2) | 85.3 (7.6) | 85.4 (7.2) | 85.3 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion
Description: Acute Insulin response during Hyperglycemic clamp (delta insulin uU/mL, t=0-10)
Time Frame: 3 hours
Population: Three subjects were excluded or withdrew after infusion but before hyperglycemic clamp due to low potassium, loss of IV access, burning at IV site. These 3 participants were not included in final analysis.
Measure: Mean (Standard Deviation); unit: uU/mL
Groups:
- Vehicle, HS: Vehicle Infusion, High Salt diet
- Vehicle, LS: Vehicle Infusion, Low Salt diet
- Aldosterone, HS: Aldosterone Infusion, High Salt diet
- Aldosterone, LS: Aldosterone Infusion, Low Salt diet
Arm/Group | Vehicle, HS | Vehicle, LS | Aldosterone, HS | Aldosterone, LS
Number analyzed (Participants) | 17 | 12 | 17 | 12
uU/mL | 48.9 (34.8) | 37.6 (30.9) | 51.8 (40.2) | 34.4 (20.9)

2. Secondary Outcome: Insulin Sensitivity
Description: Insulin sensitivity index (ISI) was calculated by dividing the average glucose infusion rate (mg glucose infusion/kg body weight/min) by the average insulin concentration (uU/mL) from 90 to 120 minutes. This was multiplied by 100 (thus, x100 in units description), per reporting convention in literature.
Time Frame: 3 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/kg/min per uU/mL*100
Arm/Group | Vehicle, HS | Vehicle, LS | Aldosterone, HS | Aldosterone, LS
Number analyzed (Participants) | 17 | 12 | 17 | 12
mg/kg/min per uU/mL*100 | 25.2 (15.4) | 24.8 (16.4) | 23.4 (17.3) | 24.7 (13.4)

ADVERSE EVENTS:
Arm/Group | Vehicle, HS | Vehicle, LS | Aldosterone, HS | Aldosterone, LS
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/14 | 0/18 | 0/14
Other Adverse Events (participants affected / at risk) | 5/18 | 4/14 | 3/18 | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle, HS (N=18) | Vehicle, LS (N=14) | Aldosterone, HS (N=18) | Aldosterone, LS (N=14)
Low potassium (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
IV site discomfort (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lightheadedness (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — during study diet, prior to drug infusion
Nasal congestion or rhinorrhea (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No